CLINICAL TRIAL: NCT03803423
Title: Dissemination of the Donor Application: Utilizing Social Media to Identify Potential Live Organ Donors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: MaineHealth (Other); Washington University School of Medicine (Other); Scripps Health (Other); Yale University (Other); Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00146922
Record Dates: First submitted 2019-01-09; First posted 2019-01-14 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: End Stage Renal Disease; End Stage Liver Disease
Keywords: Live Donor Transplant; Social Media; Advocacy; Education; Living Donation; The Donor App
MeSH Terms: conditions — Kidney Failure, Chronic; End Stage Liver Disease

STUDY DESIGN:
Intervention Model Description: All participants will be invited to use the Donor App.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The Donor App (Experimental): Select physicians and research staff from about 15 transplant hospitals will be given access to distribute the application to patients who the above people feel could benefit from the application. After obtaining informed consent, an approved member of the study team will enter the participant's name, contact info, and organ needed into the Donor App's secure management portal to send an email or text message with a unique and protected invitation link to the participant. Using this link the participant will be allowed to use the Donor App indefinitely.
  Interventions: Other: The Donor App

INTERVENTIONS:
Other: The Donor App — The Donor app is a web-based application that helps transplant candidates tell the candidate's story via social media in the hopes of identifying an appropriate living donor. Sample stories created using the Donor App can be found at www.thedonorapp.com.

SUMMARY:
This study utilizes a web-based application to help patients on the organ transplant waitlist communicate patient's need for a living donor via social media and provide interested potential donors the opportunity to engage with the evaluation process.

DETAILED DESCRIPTION:
Barriers to identifying a live donor include lack of education and hesitance to initiate a conversation about live donation. For these reasons, many transplant candidates are hesitant to discuss candidate's illness and are therefore reluctant to pursue live donor transplantation. The investigators hypothesize that utilization of social media to spread awareness about candidate's illness and candidate's need for a live donor will enable many transplant candidates to successfully identify live donors. In this study, participants will use a novel web-based application, called the "Donor App", to create and share candidate's story via Facebook and other social networks to assist in the search for a live donor.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* On the kidney-only or liver-only transplant waiting list at a collaborating center

Exclusion Criteria:

* Younger than 18 years of age
* Not on the kidney or liver transplant waiting list
* On multiple organ transplant waiting lists

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2017-11-27 (Actual); Primary Completion 2026-11-27 (Estimated); Study Completion 2026-11-27 (Estimated)

PRIMARY OUTCOMES:
Potential donors identified | Up to 5 years
  Number of potential live donors that come forward to the transplant center on behalf of the participant.
Live donor transplantation | Up to 5 years
  Number of participants that receive a live donor transplant.

SECONDARY OUTCOMES:
App utilization as assessed by number of participants with story completion and posting in the donor app | Up to 5 years
  The extent of a participants story completion and posting will be recorded internally by the Donor App. The number of participants that complete stories and post will be counted to assess app utilization.
The Donor App Implementation | Up to 5 years
  Success of the Donor App across multiple institutions will be tracked by the number of participants enrolled and invited to use the app at each institution.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Cameron, MD PhD, Principal Investigator — Johns Hopkins University
Locations (6):
- United States (6):
  - Scripps Green Hospital, San Diego, California
  - Yale University, New Haven, Connecticut
  - Rush University Medical Center, Chicago, Illinois
  - Maine Medical Center, Portland, Maine
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Washington University in St. Louis, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar K, King EA, Muzaale AD, Konel JM, Bramstedt KA, Massie AB, Segev DL, Cameron AM. A Smartphone App for Increasing Live Organ Donation. Am J Transplant. 2016 Dec;16(12):3548-3553. doi: 10.1111/ajt.13961. Epub 2016 Aug 10. PMID 27402293
- [Background] Bramstedt KA, Cameron AM. Beyond the Billboard: The Facebook-Based Application, Donor, and Its Guided Approach to Facilitating Living Organ Donation. Am J Transplant. 2017 Feb;17(2):336-340. doi: 10.1111/ajt.14004. Epub 2016 Sep 7. PMID 27501516
- See also: The Donor App Homepage — https://www.thedonorapp.com/